CLINICAL TRIAL: NCT00876772
Title: Randomized, Placebo-controlled Parallel Group Study for the Evaluation of an Oral Dose of 10mg Olanzapine in Combination With Riluzole for the Treatment of Loss of Appetite in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Olanzapine for the Treatment of Appetite Loss in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Thomas Meyer, MD, Prof. Dr. Thomas Meyer, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLN-ALS01
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; olanazapine; Loss of Apptetite; Appetite Loss; Malnutrition; Cachexia; Zyprexa
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Anorexia; Malnutrition; Cachexia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Olanzapine — Randomized, placebo-controlled, parallel group trial to evaluate the effectiveness and tolerability of an oral dose of 10 mg Olanzapine in combination with Riluzole for the treatment of Loss of Appetite in patients with amyotrophic lateral sclerosis (ALS)

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is an adult neurodegenerative disease that is caused by a selective degeneration of the motor nerve cells in the cortex and myelon. As a result of motor neurodegeneration, a progredient paralysis of the extremities and of the speaking, swallowing, and breathing musculature develops. ALS leads to death by respiratory insufficiency in a mean course of 3-5 years. More than 80% of ALS patients present with a clinically significant and undesirable weight loss. The cause of weight loss is heterogeneous. Fundamentally, the investigators must distinguish malnutrition, cachexia and loss of appetite. Loss of weight is an independent prognosis factor in ALS. Effective treatment of undesirable weight loss is an important therapy goal for ALS.

The researchers propose an investigational therapy of ALS with oral administration of Olanzapine. The rationale for this study is based on the weight-increasing effect of OLN. The clinical trial aims to employ OLN-induced weight gain or weight stabilization as a symptomatic therapy for the loss of appetite. An undesired weight loss of at least 10% of the body weight should be reduced through the weight-increasing effect of OLN. The hypothesis states that the undesired weight loss in ALS patients during treatment with OLN 10mg in combination with Riluzole (RIL) 100mg is at least 20 percentage points less than for treatment with placebo in combination with 100 mg RIL.

DETAILED DESCRIPTION:
After randomization, there is a placebo-controlled parallel group treatment with 10 mg OLN in combination with the standard treatment of Riluzole (100mg/day)(Group 1) in comparison to treatment with placebo in combination with 100 mg RIL (Group 2). Study drug will be provided as 5 mg tablets. OLN will be begun in an initial dosage of 5 mg/day for one week. The intake will occur in the evening hours in the form of a capsule containing 5 mg OLN. The evening dose of Riluzole can be taken together with the OLN medication. After one week (day 8), the dose will be increase to 10 mg OLN/day, which will be taken in the form of two capsules at the same timepoint in the evening hours. This dose will be continued for 51 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 years old
* Clinical diagnosis of definitive, probable, and possible ALS (revised El Escorial Criteria) or diagnosis of the clinical ALS-variants of Progressive Muscle Atrophy (PMA)
* Sporadic and familial ALS
* Beginning of symptoms of paralysis at least 6 months prior
* Treatment with a steady dose of RIL 100 mg/day for at least 1 month
* A score of ≤ 28 in the symptom-oriented Council on Nutrition appetite questionnaire (CNAQ) by which appetite is evaluated
* Patient consent

Exclusion Criteria:

* Patients with known hypersensitivity to OLN, RIL, or one of the active ingredients
* Percutaneous Endoscopic Gastronomy (PEG)
* Clinically significant eating disorder
* Deliberate weight loss
* Underlying consumptive disease with undesired weight loss
* Overweight with BMI ≥ 25 kg/m2
* Clinically significant hypotonia and history of recurrent syncopes (> 1 syncope)
* Clinically severe concomitant illnesses, including psychiatric illnesses
* Pregnant or nursing women
* Severe neutropenia (< 750/mm3)
* Open angle glaucoma
* Diabetes mellitus
* Prostatic hyperplasia
* Extrapyramidal movement disorders including from late dyskinesia
* Dementia and incompetence to grant informed consent
* Clinically significant EKG changes
* EKG proof of a QT time corrected according to Fridericia (QTcF) > 500 ms
* Treatment with substances that are metabolized by the Cytochrom-P450-System CYP1A2 (e. g. Carbamazepine, Fluvoxamin, and Ciprofloxacin)
* Treatment with Mirtazapine within the past 3 months
* Treatment with steroids or appetite-stimulating substances including anabolics within the past 3 months
* Treatment with Valproat within the past 3 months
* Treatment with hepatotoxic medicines
* Treatment with tetrahydrocannabinol within the past 3 months
* Treatment with another atypical or typical neuroleptic within the past 3 months
* Treatment with any other study medication < 1 month before the beginning of the study
* Destructive use of psychotropic substances within the past 3 months
* Destructive use of alcohol
* Laboratory parameters outside the normal range that are associated with a clinically significant cardiovascular, pulmonologic, hematologic, hepatological, metabolic, or renal disease or that interfere with interpretation of the clinical study or that require medications that are not permitted in the study protocol
* Elevation of the serum transaminase levels (ALT/AST) to more than 3-times of the upper normal value
* Elevation of the bilirubin and gamma glutamyl transferase levels (GGT) to beyond the maximum normal value
* History of a cardiopulmonary reanimation und prevention of sudden cardiac death
* History of clinically significant EKG changes
* History of thrombotic events including deep leg vein thrombosis and pulmonary artery embolism
* History of a paralytic ileus
* History of epilepsy or an episodic seizure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Self-evaluation of appetite by using the Council on Nutrition appetite questionnaire (CNAQ) | 1 month

SECONDARY OUTCOMES:
Number and severity of adverse events (AE) and severe adverse events (SAE) | 1 month
Number of patients who have completed treatment with OLN in combination with RIL in comparison with placebo treatment in combination with RIL | 1 month
Body Mass Index (BMI) measured in body weight [kg]/(body length [m])2 | 1 month
Number of patients with a BMI <18.5 kg/m2 | 1 month
Median daily oral food intake in [kcal] which will be determined retrospectively and anamnestically by composing a dietary protocol and by conducting a standardized interview | 1 month
Median daily energy balance [kcal] (difference between actual food intake and target food intake)determined retrospectively and anamnestically by composing a dietary protocol and by conducting a standardized interview | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, MD, Principal Investigator — Charité University Hospital, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin, Berlin, Germany, Berlin, Germany